CLINICAL TRIAL: NCT02763722
Title: Evaluating Results of Regularly Applied Emollient - Spray in Atopic Dermatitis Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Wojciech Feleszko, MD PhD, Medical University of Warsaw
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB/4/2016
Record Dates: First submitted 2016-04-25; First posted 2016-05-05 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-06

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; allergic contact dermatitis; cosmetics; transepidermal water loos
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis, Allergic Contact

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Emollient spray product (Experimental): Study design
  A 3 visits are planned:
  0 week (first visit) 2nd week (second visit) 4th week (third visit)
  B. During each visit will be made:
  1. The clinical examination (including an assessment of any adverse effects)
  2. Evaluation of transepidermal water loss (TEWL) and capacitance of outer areas of the stratum corneum as an indirect assessment of skin hydration,
  3. fill out questionnaires CDLQI (The Children's Dermatology Life Quality Index)
  4. will assess VAS (visual analogue scale)
  C. All patients will be instructed to use emollients spray the entire surface of the skin at least twice daily for four weeks.
  Interventions: Other: Emollient spray product

INTERVENTIONS:
Other: Emollient spray product — All patients will be instructed to use emollients spray on entire skin at least twice a day for four weeks.
  Other Names: Atopic deramtitis group

SUMMARY:
Atopic dermatitis (AD) is a chronic, relapsing, inflammatory skin disease that has potential for profound and far-reaching effects on all aspects of children and their families lives, significantly reducing the quality of life. Atopic dermatitis typically appears in infancy and nowadays is affecting up to 10-30% of children and 2-10% of adults.

Diminished skin barrier is the essential factor that plays a role in the initiation, consolidating and exacerbating AD. Treatment options for AD typically address skin barrier protection or inflammatory components of disease. Proper care using mild and appropriately formulated emollient preparations may provide significant benefits.

In investigators prior study, more than half of pharmacy-derived emollient preparations contained potential contact haptens listed in the European baseline series (EBS), used in diagnosing contact dermatitis.

The primary aim of this study is to demonstrate the efficacy of regularly applied emollient in an atomiser (in the form of oil-in-water emulsion) in maintenance therapy, in children presenting from mild to moderate atopic dermatitis.

In this study 3 visits are planned (for a period of 4 weeks). During each visit investigators will evaluate transepidermal water loss (TEWL), capacitance of outer areas of the stratum corneum as an indirect assessment of skin hydration. Moreover, investigators will assess three-them-severityIndex and the Children's Dermatology Life Quality Index (CDLQI).

The product that participants will use in the study, was prepared at investigators request, in collaboration with the cosmetics company, which according to investigators knowledge at present, will not be benefited from the audit. The following described study project (prospective clinical trial, uncontrolled, open-label) will be conducted within the framework of the statutory tasks of the Department of Pulmonology and Allergology of Children Medical University of Warsaw and is a non-commercial project.

DETAILED DESCRIPTION:
Atopic dermatitis (AD) is a chronic, relapsing, inflammatory skin disease that has potential for profound and far-reaching effects on all aspects of children and their families lives, significantly reducing the quality of life. Atopic dermatitis typically appears in infancy and nowadays is affecting up to 10-30% of children and 2-10% of adults.

Diminished skin barrier is the essential factor that plays a role in the initiation, consolidating and exacerbating AD. The skin exposed to aeroallergens (pollen, pet dander, dust mites), or food allergens (eggs, milk, wheat protein, chocolate, strawberry), hard water, and soaps and detergents, loses the protective barrier composed of lipids (ie. Lipid) and becomes the victim of harmful, exogenous substances.

The main symptoms of atopic dermatitis are redness and dry skin, itching, moreover patients are susceptible to recurrent superficial skin infections. Skin lesions in AD are mostly located on the elbows and knees, face and neck, however they can spans the entire body. Treatment options for AD typically address skin barrier protection or inflammatory components of disease. Proper care using mild and appropriately formulated emollient preparations may provide significant benefits.

Previous observations indicated to be reasonable to selection carefully composition of emollient preparations. In investigators prior study, more than half of emollient preparations, available in online drugstores, contained potential contact sensitizers, included to 28, the most common, haptens listed in the European baseline series (EBS), used in diagnosing contact dermatitis. A significant number of investigated products contained at least two different haptens which may threaten unpredictable allergic reactions in the case of concomitance of various allergens.

The primary aim of this study is to demonstrate the efficacy of regularly applied emollient in an atomiser (in the form of oil-in-water emulsion) in maintenance therapy, in children presenting from mild to moderate atopic dermatitis.

The composition of the tested emollient is typical and based on the frequently occurring substances found in public preparations of this kind.

Emollient spray (composition INCI):

Aqua, Glycerin, Aqua, Parfum, Glyceryl Caprylate, Allantoin, Xanthan Gum, Butyrospermum Parkii Butter, Adansonia digitata Seed Oil, Oenothera Biennis Oil, Perilla ocymoides Seed Oil, Tocopheryl Acetate, Palm Kernel Glycerides, Squalane, behenyl Alcohol, Glyceryl Stearate, Palmitic Acid, Stearic Acid, Lecythin, Cetyl Alcohol, Myristyl Alcohol, Ceramide NP, Glyceryl Stearate Citrate, Cetearyl Alcohol, Tocopheryl Acetate, Caprylic / Capric Trigliceride, Dicaprylyl Carbonate, Tocopherol, Etylhexyl Stearate.

The product that will be used in the study (emollients in spray- composition of the product given above) was prepared at investigators request, in collaboration with the cosmetics company, which according to investigators knowledge at present, will not be benefited from the audit.

The following described study project will be conducted within the framework of the statutory tasks of the Department of Pulmonology and Allergology of Children Medical University of Warsaw and is a non-commercial project.

ELIGIBILITY:
Inclusion Criteria:

A. Clinical diagnosis of atopic dermatitis (AD) using the criteria Hanifin and Rajka

Exclusion Criteria:

A. severe atopic dermatitis (SCORAD Index over 40) B. oral steroids dose over 1 mg / kg. eq prednisolone or other oral immunosuppressive drugs during the last 3 days C. topical steroids or calcineurin inhibitors used more than 1 week D. viral skin infection (eg. Eczema herpeticum) or bacterial infections of the skin, E. severe systemic disease (kidney failure, heart disease, immunodeficiency)

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-05; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Change from Transepidermal Water Loss (TEWL) | 4 weeks
  Standardized measurements of evaporation percutaneous (transepidermal water loss, TEWL) and capacitance outer areas of the stratum corneum giving indirect evaluation of skin hydration will be performed by the same researcher. The tests will be carried out always at the same point of the body.

SECONDARY OUTCOMES:
Change from the Children's Dermatology Life Quality Index (CDLQI ) | 4 weeks
  Courtesy of Professor A. Y. Finlay and Dr. M. S. Lewis-Jones of the Medical University of Cardiff during the study will be used a questionnaire about quality of life in children suffering from dermatological diseases.
Change from scoring atopic dermatitis index (SCORAD Index) | 4 weeks

OTHER OUTCOMES:
Change from three-item-severity indicator (TIS) | 4 weeks
  TIS evaluats the severity of erythema (max. 3 points), swelling (max. 3 points) and scratchs (max. 3 points), the maximum value of TIS = 9.

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Feleszko, MD PhD, Principal Investigator — Department of Pediatric Respiratory Diseases and Allergy, The Medical University of Warsaw
Locations (1):
- Katarzyna Osinka, Warsaw, Żwirki I Wigury 63A, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eichenfield LF, Tom WL, Berger TG, Krol A, Paller AS, Schwarzenberger K, Bergman JN, Chamlin SL, Cohen DE, Cooper KD, Cordoro KM, Davis DM, Feldman SR, Hanifin JM, Margolis DJ, Silverman RA, Simpson EL, Williams HC, Elmets CA, Block J, Harrod CG, Smith Begolka W, Sidbury R. Guidelines of care for the management of atopic dermatitis: section 2. Management and treatment of atopic dermatitis with topical therapies. J Am Acad Dermatol. 2014 Jul;71(1):116-32. doi: 10.1016/j.jaad.2014.03.023. Epub 2014 May 9. PMID 24813302
- [Background] Zukiewicz-Sobczak WA, Adamczuk P, Wroblewska P, Zwolinski J, Chmielewska-Badora J, Krasowska E, Galinska EM, Cholewa G, Piatek J, Kozlik J. Allergy to selected cosmetic ingredients. Postepy Dermatol Alergol. 2013 Oct;30(5):307-10. doi: 10.5114/pdia.2013.38360. Epub 2013 Oct 30. PMID 24353491
- See also: our prior study — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4401009/
- See also: similar method of the study project — http://www.termedia.pl/Original-papers-The-influence-of-emollient-Eucerin-174-Soothing-lotion-12-Omega-on-transepidermal-water-loss-moisturization-of-epidermis-and-skin-elasticity-in-children-with-atopic-dermatitis,7,11915,0,1.html